CLINICAL TRIAL: NCT00291577
Title: Exploratory Evaluation Of A Sequential Administration Of Docetaxel And SU011248 In Women With Advanced Breast Cancer
Brief Title: Study Of SU011248 In Combination With Docetaxel In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181100
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-11

CONDITIONS: Breast Neoplasms
Keywords: advanced; sunitinib (Sutent); docetaxel; Phase 1B
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib (Sutent); Drug: Taxotere

INTERVENTIONS:
Drug: Sunitinib (Sutent) — Sunitinib (Sutent) 37.5 mg in schedule 2/1; Sunitinib (Sutent) 37.5 mg in continuous dosing (post discontinuation of axotere) and in accordance with Investigator decision
  Other Names: Sutent
Drug: Taxotere — Taxotere 75 mg/m2 iv, once every 3 weeks

SUMMARY:
This study is to evaluate the safety of SU011248 (Sunitinib/Sutent) in combination with docetaxel in patients with metastatic or locally recurrent breast cancer who have not received chemotherapy treatment in the advanced disease setting.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with evidence of unresectable, locally recurrent or metastatic disease
* Candidate for treatment with docetaxel

Exclusion Criteria:

* Prior chemotherapy in the advanced disease setting
* Inflammatory breast cancer
* HER2 positive disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Milan, Italy
- Pfizer Investigational Site, Stockholm, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181100&StudyName=Study%20Of%20SU011248%20In%20Combination%20With%20Docetaxel%20In%20Patients%20With%20Metastatic%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First 12 subjects evaluable for pharmacokinetic (PK) analysis had full PK profile on Cycle 1, Day 1 (C1D1) and C2D1.
Groups:
- Sunitinib in Combination With Docetaxel: Sunitinib (SU011248) orally (PO) for 2 weeks every 3 weeks (2 weeks on, then 1 week off = Schedule 2/1) starting on Day 2 (Cycle 2, Day 3 only for those subjects included in the Pharmacokinetic [PK] study); starting dose 37.5 milligrams (mg) daily (QD). Docetaxel (Taxotere) administered Day 1 of each cycle via intravenous (IV) infusion every 3 weeks; starting dose 75 mg/m2.
Period: Overall Study
Arm/Group | Sunitinib in Combination With Docetaxel
Started | 22
Completed | 1 (Subject End of Study=Completed; not per protocol reason. PI reason=withdrawn during active treatment)
Not Completed | 21
Not completed — Adverse Event | 1
Not completed — Other | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 14

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 22
Age, Customized [Number; unit: participants]
  18 to 44 years | 3
  45 to 64 years | 13
  > = 65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters
Description: Median Tmax = time for maximum plasma concentration (Cmax) for SU011248, SU012662, and combined SU011248 and SU012662 (total drug); collected C1D2, C2D3. Paired observation.
Time Frame: 1, 2, 4, 6, 8, 12, 24 hours postdose
Population: Evaluable set of subjects for PK analysis is subjects in ITT population who completed sampling for PK profiles for both SU011248 and docetaxel; ITT population = all subjects enrolled in study who received at least 1 dose of study medication (SU011248 or docetaxel).
Measure: Median (Full Range); unit: hours
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 11
hours
  SU011248 C1D2 | 6.0 [4.0 to 24.0]
  SU011248 C2D3 | 6.0 [2.0 to 8.0]
  SU012662 C1D2 | 6.0 [2.0 to 24.0]
  SU012662 C2D3 | 6.0 [4.0 to 24.0]
  Total drug C1D2 | 6.0 [2.0 to 24.0]
  Total drug C2D3 | 6.0 [2.0 to 8.0]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters
Description: Mean Cmax = maximum plasma concentration for SU011248, SU012662, and combined SU011248 and SU012662 (total drug) measured as nanograms per milliliter (ng/mL); collected C1D2, C2D3. Paired observation; Cmax dose corrected C2D3 (dose correction if predose concentrations of SU011248 or SU012662 were > 5% of Cmax).
Time Frame: 1, 2, 4, 6, 8, 12, 24 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 11
ng/mL
  SU011248 C1D2 | 29.17 (7.906)
  SU011248 C2D3 | 29.49 (7.910)
  SU012662 C1D2 | 5.07 (2.385)
  SU012662 C2D3 | 5.91 (2.251)
  Total drug C1D2 | 34.05 (9.312)
  Total drug C2D3 | 34.69 (8.941)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; SU011248 C1D2 vs C2D3. Due to the exploratory nature of the study, no statistical hypothesis testing was done since the primary purpose was to assess the tolerability of the combination of SU011248 with docetaxel; Test type: Superiority or Other; Ratio of adjusted geometric means = 98.89, 90% CI [80.34 to 121.73] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale
Statistical Analysis 2: Comparison: Sunitinib in Combination With Docetaxel; SU012662 C1D2 vs C2D3; Test type: Superiority or Other; Ratio of adjusted geometric means = 81.96, 90% CI [59.76 to 112.41] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale
Statistical Analysis 3: Comparison: Sunitinib in Combination With Docetaxel; Total drug C1D2 vs C2D3; Test type: Superiority or Other; Ratio of adjusted geometric means = 97.81, 90% CI [80.44 to 118.94] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

3. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero (0) to 24 Hours (AUC24): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters
Description: Mean AUC24 = area under plasma concentration-time profile from time 0 to 24 hours for SU011248, SU012662, and combined SU011248 and SU012662 (total drug) measured in nanograms times hour per milliliter (ng*hr/mL); collected C1D2, C2D3. Paired observation; AUC24 dose corrected C2D3 (dose correction if predose concentrations of SU011248 or SU012662 were > 5% of Cmax).
Time Frame: 1, 2, 4, 6, 8, 12, 24 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 11
ng*hr/mL
  SU011248 C1D2 | 486.38 (132.439)
  SU011248 C2D3 | 479.80 (128.718)
  SU012662 C1D2 | 82.21 (33.204)
  SU012662 C2D3 | 96.88 (30.513)
  Total drug C1D2 | 568.78 (152.106)
  Total drug C2D3 | 567.43 (145.952)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; SU011248 C1D2 vs C2D3; Test type: Superiority or Other; Ratio of adjusted geometric means = 101.23, 90% CI [82.75 to 123.83] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale
Statistical Analysis 2: Comparison: Sunitinib in Combination With Docetaxel; SU012662 C1D2 vs C2D3; Test type: Superiority or Other; Ratio of adjusted geometric means = 81.72, 90% CI [62.40 to 107.04] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale
Statistical Analysis 3: Comparison: Sunitinib in Combination With Docetaxel; Total drug C1D2 vs C2D3; Test type: Superiority or Other; Ratio of adjusted geometric means = 100.00, 90% CI [82.95 to 120.56] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

4. Primary Outcome: Area Under the Curve From Time 0 to Last Quantifiable Concentration (AUClast): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters
Description: Mean AUClast = area under the plasma concentration-time profile from time 0 (predose) to the last measurable concentration; collected C1D2, C2D3. Data did not allow calculation of AUClast; not summarized; AUC summarized in outcome measure: Area under the plasma concentration-time curve from time zero (0) to 24 hours (AUC24): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters.
Time Frame: 1, 2, 4, 6, 8, 12, 24 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 0

5. Primary Outcome: Trough Plasma Concentration (Ctrough) at Time Zero (0): Sunitinib (SU011248), Sunitinib Metabolite (SU012662), and Total Drug PK Parameters
Description: Mean Ctrough=plasma concentration-time profile at time 0 (predose); collected C1D2, C1D15, and C2D1. Calculated by setting concentration values below the limit of quantification to zero.
Time Frame: 0 hour postdose
Population: Evaluable set of subjects for PK analysis; (n) = Number of observations above lower limit of quantification (NALQ). No participants analyzed for SU011248 C1D2 and SU012662 C1D2; standard deviation for Total drug C1D2 confirmed as 0.00 (median, minimum, and maximum = 0.20).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 18
ng/mL
  SU011248 C1D15 (n=18) | 52.06 (23.05)
  SU011248 C2D1 (n=11) | 5.00 (5.14)
  SU012662 C1D15 (n=18) | 21.75 (8.85)
  SU012662 C2D1 (n=11) | 4.88 (3.52)
  Total drug C1D2 (n=12) | 0.20 (0.00)
  Total drug C1D15 (n=18) | 73.81 (29.00)
  Total drug 21D1 (n=11) | 9.87 (8.36)

6. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax): Docetaxel PK Parameters
Description: Median Tmax = time to maximum plasma concentration (Cmax) for Docetaxel; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Median (Full Range); unit: hours
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
hours
  C1D1 | 0.70 [0.5 to 1.0]
  C2D1 | 0.77 [0.5 to 1.0]

7. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Docetaxel PK Parameters
Description: Mean Cmax = maximum plasma concentration for Docetaxel; collected C1D1, C2D1. Paired observation; Cmax dose corrected (dose correction if predose concentrations of SU011248 or SU012662 were > 5% of Cmax).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
ng/mL
  C1D1 | 2932.00 (903.952)
  C2D1 | 2955.38 (853.925)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; C1D1 vs C2D1; Test type: Superiority or Other; Ratio of adjusted geometric means = 99.18, 90% CI [78.73 to 124.95] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (0) to 24 Hours (AUC24): Docetaxel PK Parameters
Description: Mean AUC24 = area under the plasma concentration-time profile from time 0 to 24 hours; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
ng*hr/mL
  C1D1 | 2918.09 (594.227)
  C2D1 | 3101.69 (778.041)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; C1D1 vs C2D1; Test type: Superiority or Other; Ratio of adjusted geometric means = 94.98, 90% CI [78.73 to 114.58] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

9. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment
Description: Median time (50 percent [%]) from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first; based on Investigator assessment. PFS calculated as (Weeks) = (first event date minus first dose date plus 1) divided by 7.
Time Frame: First dose of study treatment until progressive disease
Population: ITT population = all subjects enrolled in study who received at least 1 dose of study medication (SU011248 or docetaxel).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 20
weeks | 34.9 [28.1 to 55.6]

10. Secondary Outcome: Number of Subjects With Objective Response of Complete Response or Partial Response Based on Investigator Assessment
Description: Number of subjects with objective response based on Investigator assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
Time Frame: First dose of study treatment until at least 4 weeks after confirmed response or partial response
Population: ITT; subjects with baseline assessments
Measure: Number; unit: participants
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 20
participants | 14 [lower limit 90.9]
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; Overall confirmed objective response rate (CR + PR); Test type: Superiority or Other; rate (percent) = 73.7, 95% CI [48.8 to 90.9] — Two-sided Confidence Interval (CI) (%) from exact method based on F distribution

11. Secondary Outcome: Number of Subjects With Clinical Benefit of Complete Response, Partial Response, or Stable Disease Based on Investigator Assessment
Description: Number of subjects with clinical benefit based on Investigator assessment of confirmed complete response (CR), partial response (PR), or stable disease (SD) according to RECIST for at least 24 weeks on study.
Time Frame: First dose of study treatment until at least 24 weeks on study
Population: ITT; subjects with baseline assessments
Measure: Number; unit: participants
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 20
participants | 17
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; Clinical Benefit Rate (CR + PR + SD > = 24 weeks); Test type: Superiority or Other; rate (percent) = 89.5, 95% CI [66.9 to 98.7] — Two-sided CI (%) from exact method based on F distribution

12. Secondary Outcome: Duration of Tumor Response Based on Investigator Assessment
Description: Median duration (50%) of tumor response based on Investigator assessment for a subgroup of subjects with objective disease response: who have not progressed or died due to any cause; with a response and subsequent progression or death due to any cause for duration of response (DR). DR defined as time from start of first documented objective tumor response (CR or PR) to first documented objective tumor progression or death due to any cause, whichever occurs first. DR calculated as (Weeks) = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.
Time Frame: Start of first confirmed CR or PR to first confirmed progression or death
Population: ITT; subgroup of subjects with objective disease response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 14
weeks | 28.7 [22.7 to 69.6]

13. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (0) to 48 Hours (AUC48): Docetaxel PK Parameters
Description: Mean AUC48 = area under the plasma concentration-time profile from time 0 to 48 hours; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr.mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
ng*hr.mL
  C1D1 | 3167.53 (658.124)
  C2D1 | 3326.98 (775.599)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; C1D1 vs C2D1; Test type: Superiority or Other; Ratio of adjusted geometric means = 95.57, 90% CI [79.90 to 114.32] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

14. Primary Outcome: Area Under the Curve From Time 24 Hours to 48 Hours (AUC24_48) : Docetaxel PK Parameters
Description: Mean AUC24_48 = area under the plasma concentration-time profile from 24 to 48 hours; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
ng*hr/mL
  C1D1 | 249.45 (108.911)
  C2D1 | 225.29 (96.657)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; C1D1 vs C2D1; Test type: Superiority or Other; Ratio of adjusted geometric means = 112.39, 90% CI [81.05 to 155.85] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

15. Primary Outcome: Area Under the Curve From Time 0 to Last Quantifiable Concentration (AUClast): Docetaxel PK Parameters
Description: Mean AUClast = area under the plasma concentration-time profile from time 0 (predose) to the last measurable concentration; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 10
ng*hr/mL
  C1D1 | 3159.58 (675.834)
  C2D1 | 3304.48 (769.011)
Statistical Analysis 1: Comparison: Sunitinib in Combination With Docetaxel; C1D1 vs C2D1; Test type: Superiority or Other; Ratio of adjusted geometric means = 95.79, 90% CI [79.82 to 114.96] — Ratio percent (%) (Test/Reference) of adjusted geometric means; values have been back-transformed from the log scale

16. Primary Outcome: Plasma Elimination Half-life (t1/2): Docetaxel PK Parameters
Description: Mean Thalf (t1/2) = terminal elimination half life; collected C1D1, C2D1. Paired observation.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 32, 48 hours postdose
Population: Evaluable set of subjects for PK analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sunitinib in Combination With Docetaxel
Number analyzed (Participants) | 9
hours
  C1D1 | 22.55 (5.914)
  C2D1 | 24.88 (10.651)

ADVERSE EVENTS:
Arm/Group | Sunitinib in Combination With Docetaxel
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib in Combination With Docetaxel (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib in Combination With Docetaxel (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 10
Conjunctivitis (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 3
Photopsia (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 7
Glossodynia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Oral pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 6
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 4
Face oedema (General disorders) | 2
Fatigue (General disorders) | 10
Local swelling (General disorders) | 2
Mucosal inflammation (General disorders) | 9
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 3
Pyrexia (General disorders) | 7
Cystitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 6
Alanine aminotransferase (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 8
Paraesthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other